CLINICAL TRIAL: NCT06525883
Title: Analysis of Patients With Post-traumatic Vertebral Fracture and Accompanying Rib Fracture
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Gizem Kececi Ozgur, Principal investigator, Ege University
Other Study IDs: 2023-0312
Record Dates: First submitted 2024-07-25; First posted 2024-07-29 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Vertebral Fracture; Rib Fractures; Trauma
Keywords: trauma; rib fracture; vertebral fracture; complication
MeSH Terms: conditions — Spinal Fractures; Rib Fractures; Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: upper cervical
  Interventions: Other: No intervation
- Group 2: lower cervical
  Interventions: Other: No intervation
- Group 3: thoracolumbar
  Interventions: Other: No intervation

INTERVENTIONS:
Other: No intervation — No intervention was made to the groups

SUMMARY:
The present study investigates the trauma mechanisms, the type and level of vertebral fractures, the number of accompanying rib fractures and thoracic pathologies, the surgical procedures employed and the development of complications in a sample of patients who presented with vertebral fractures and concurrent rib fractures after sustaining trauma.

DETAILED DESCRIPTION:
The study aimed to analyze the mechanisms of trauma, type and level of vertebral fractures, number of accompanying rib fractures and thoracic pathologies, necessity of surgery and development of complications in patients who developed vertebral fractures and rib fractures after trauma. Patients were divided into 3 groups: upper cervical , lower cervical and thoracolumbar. They were compared with each other in terms of trauma mechanisms, rib fracture numbers, accompanying thoracic pathologies, complication developments and need for surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had vertebral and rib fractures due to trauma

Exclusion Criteria:

* Patients whose electronic patient records and radiological imaging findings cannot be accessed
* Patients whose development of complications could not be evaluated due to not coming to post-discharge check-ups

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who had vertebral and rib fractures due to trauma
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
rib fracture | 12 months
  number of accompanying rib fractures
complications | 12 months
  Number of patients developing complications
surgical intervention | 12 months
  Number of patients requiring surgical intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University Faculty of Medicine, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The dataset of the research presented in this article is under record. Corresponding author can be contacted to reach the required data network.

REFERENCES:
- [Result] Broderick SR. Hemothorax: Etiology, diagnosis, and management. Thorac Surg Clin. 2013 Feb;23(1):89-96, vi-vii. doi: 10.1016/j.thorsurg.2012.10.003. Epub 2012 Nov 3. PMID 23206720
- [Result] Cameron P, Dziukas L, Hadj A, Clark P, Hooper S. Rib fractures in major trauma. Aust N Z J Surg. 1996 Aug;66(8):530-4. doi: 10.1111/j.1445-2197.1996.tb00803.x. PMID 8712986
- [Result] Coary R, Skerritt C, Carey A, Rudd S, Shipway D. New horizons in rib fracture management in the older adult. Age Ageing. 2020 Feb 27;49(2):161-167. doi: 10.1093/ageing/afz157. PMID 31858117
- [Result] Looby S, Flanders A. Spine trauma. Radiol Clin North Am. 2011 Jan;49(1):129-63. doi: 10.1016/j.rcl.2010.07.019. PMID 21111133
- [Result] Ahern DP, McDonnell J, O Doinn T, Butler JS. Timing of surgical fixation in traumatic spinal fractures: A systematic review. Surgeon. 2020 Feb;18(1):37-43. doi: 10.1016/j.surge.2019.04.002. Epub 2019 May 4. PMID 31064710
- [Result] Yang Z, Lowe AJ, de la Harpe DE, Richardson MD. Factors that predict poor outcomes in patients with traumatic vertebral body fractures. Injury. 2010 Feb;41(2):226-30. doi: 10.1016/j.injury.2009.10.019. Epub 2009 Nov 3. PMID 19889411
- [Result] Chiu WT, Lin HC, Lam C, Chu SF, Chiang YH, Tsai SH. Review paper: epidemiology of traumatic spinal cord injury: comparisons between developed and developing countries. Asia Pac J Public Health. 2010 Jan;22(1):9-18. doi: 10.1177/1010539509355470. PMID 20032030
- [Result] Aghakhani K, Kordrostami R, Memarian A, Asl ND, Zavareh FN. The association between type of spine fracture and the mechanism of trauma: A useful tool for identifying mechanism of trauma on legal medicine field. J Forensic Leg Med. 2018 May;56:80-82. doi: 10.1016/j.jflm.2018.01.004. Epub 2018 Feb 7. PMID 29571167
- [Result] Oken F, Yildirim O, Oken O, Gulcek M, Yavuzer G, Ucaner A. Short or long fusion after thoracolumbar burst fractures does not alter selected gait parameters: a preliminary study. J Orthop Res. 2011 Jun;29(6):915-8. doi: 10.1002/jor.21329. Epub 2011 Jan 21. PMID 21259336
- [Result] Machino M, Yukawa Y, Ito K, Nakashima H, Kato F. Posterior/anterior combined surgery for thoracolumbar burst fractures--posterior instrumentation with pedicle screws and laminar hooks, anterior decompression and strut grafting. Spinal Cord. 2011 Apr;49(4):573-9. doi: 10.1038/sc.2010.159. Epub 2010 Nov 16. PMID 21079623
- [Result] Wang H, Zhang Y, Xiang Q, Wang X, Li C, Xiong H, Zhou Y. Epidemiology of traumatic spinal fractures: experience from medical university-affiliated hospitals in Chongqing, China, 2001-2010. J Neurosurg Spine. 2012 Nov;17(5):459-68. doi: 10.3171/2012.8.SPINE111003. Epub 2012 Sep 14. PMID 22978439
- [Result] Watanabe M, Sakai D, Yamamoto Y, Sato M, Mochida J. Upper cervical spine injuries: age-specific clinical features. J Orthop Sci. 2010 Jul;15(4):485-92. doi: 10.1007/s00776-010-1493-x. Epub 2010 Aug 19. PMID 20721716
- [Result] Rosenthal BD, Boody BS, Jenkins TJ, Hsu WK, Patel AA, Savage JW. Thoracolumbar Burst Fractures. Clin Spine Surg. 2018 May;31(4):143-151. doi: 10.1097/BSD.0000000000000634. PMID 29578877
- See also: Türkiye İstatistik Kurumu (TUİK). Ölüm ve Ölüm Nedeni İstatistikleri, 2019. — https://data.tuik.gov.tr/Bulten/Index?p=Olum-ve-Olum-Nedeni-Istatistikleri-2019-33710